CLINICAL TRIAL: NCT05761769
Title: Twin Pregnancy: a Challenge for Patients, Families and Health Professionals
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3797
Record Dates: First submitted 2023-02-13; First posted 2023-03-09 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Twin Pregnancy With Antenatal Problem; Twin Diseases; Twin Placenta
MeSH Terms: conditions — Diseases in Twins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Twin pregnancies represent 3-4% of all births and in the last two decades the rate of twin pregnancies has steadily increased, essentially due to the spread of assisted fertilization techniques, the use of drugs that stimulate ovulation and increase in maternal age at conception.

Multiple pregnancies pose unique challenges for the patient, families, caregivers and society. Indeed, twin pregnancy is associated with an increased risk compared with singleton pregnancies of all feto-maternal complications of pregnancy (Level of Evidence II-2).

In twin pregnancies (both monochorionic, MC, and bichorionic, BC) the incidence of preeclampsia is about 10%, 3 times higher than in singleton pregnancies. In singleton pregnancy, the mean gestational age (GE) at delivery is 39 weeks, the mean GA at delivery in twin pregnancies is less than 36 weeks, reflecting a 9-fold higher prevalence of spontaneous preterm delivery than in singleton pregnancy. Gestational diabetes complicates about 22% of twin pregnancies compared to 7-11% of singleton pregnancies. Twin pregnancy, compared to single pregnancy, has an increased incidence of perinatal and neonatal mortality, low birth weight, chromosomal or structural defects.

A key factor to know is chorionicity. Chorionicity is a key data to acquire in the first trimester. Indeed, some complications of twin pregnancy are specific to MC pregnancy. About 20-33% of twins share the same placenta and it is precisely in these cases that a condition of greater risk is created. The most common complications of MC pregnancy are: twin-to-twin transfusion syndrome (TTTS), due to the presence of vascular anastomoses at the level of the placenta and a clear imbalance in blood flow between the twins; selective intrauterine growth restriction; the anemia-polycythemia sequence (TAPS); twin reversed arterial perfusion (TRAPS). Thus, the MC twin pregnancy is at increased risk of feto-maternal complications.

The complications of twin pregnancy place a heavy emotional and economic burden on parents, families and society.

There is no consensus in the literature on what should be the most appropriate methods for surveillance of multiple pregnancy: when to perform laboratory, instrumental and diagnostic tests for follow-up and monitoring of maternal-fetal well-being.

The aim of this project is to create a complete and accurate database that takes into consideration all aspects related to twin pregnancy. The twin pregnancy will be followed by a team of multiple pregnancy specialists who will follow the international guidelines for the surveillance of multiple pregnancy. The aim is to identify the optimal management of multiple pregnancy, collecting, studying and comparing the largest possible number of clinical, laboratory and ultrasound data from the beginning of pregnancy to the postpartum visit, developing clinical-diagnostic care pathways for follow-up and possible prevention of complications, personalized and adapted to each single woman with a twin pregnancy.

The women participating in the study will be able to enjoy close surveillance by a center specialized in the management of multiple pregnancies, this will allow for optimal management of the twin pregnancy with early identification and treatment of any complications identified.

Study typology Prospective observational longitudinal study of the overall management of patients with multiple pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > 18 years
* Twin pregnancy with two or more viable fetuses
* Signature of the informed consent

Exclusion Criteria:

* Women without the ability to understand the protocol
* Women for whom the attending physician contraindicates participation in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women with BC or MC twin pregnancies, who arrive, consecutively, in our Multiple Pregnancy Clinic, at the Obstetrics Day Hospital, regardless of gestational age, will be invited to participate in the project
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the outcomes between twin pregnancies with and without complications after introducing a specific clinical surveillance protocol that complies with the international guidelines available. | through study completion, an average of 1 year
  To compare the outcomes between twin pregnancies with and without complications after introducing a specific clinical surveillance protocol that complies with the international guidelines available.
Identify the optimal management of multiple pregnancy, identifying markers or combination of biomarkers for the early prevention of complications in multiple pregnancy in the first, second or third trimester | through study completion, an average of 1 year
  Identify the optimal management of multiple pregnancy, identifying markers or combination of biomarkers for the early prevention of complications in multiple pregnancy in the first, second or third trimester

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Bevilacqua, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code